CLINICAL TRIAL: NCT04424173
Title: The Effect of Low Dose Combined Hormone Therapy (Estradiol And Norethindrone Acetate) on Serum CRP Levels and Life Quality in Natural Menopause Women
Brief Title: Combined Hormone Therapy, C-reactive Protein(CRP) Levels and Life Quality in Natural Menopause Women
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, professor, Karadeniz Technical University
Other Study IDs: 2007/25
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: CRP; Menopause
Keywords: CRP; Estradiol; Menopause-Specific Quality of Life questionnaire; Norethindrone Acetate.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the effect of low dose combined estradiol and norethindrone acetate hormone therapy on serum CRP levels and life quality in natural menopause women. 45 natural menopause women who admitted to Karadeniz Technical University, Faculty of Medicine, Department of Obstetrics and Gynaecology for 1 year and diagnosed as menopause and planned to have hormone therapy for menopausal symptoms involved in this study. The serum CRP levels and vasomotor symptoms scores graded according to Blatt-Kupperman Index and life quality scores according to Menopause-Specific Quality of Life Questionnaire (MENQOL) in Turkish were recorded before and after (3 months later) low dose hormone treatment (1 mg Estradiol and 0.5 mg Norethindrone acetate).

ELIGIBILITY:
Inclusion Criteria:

* Accepting consent to participate in the research and signing the form;
* Postmenopausal women 45-55 years old
* not having had menstruation for the past 6 months;
* Hormone results compatible with menopause (FSH> 20 milli-International unit(mIU) / mL, E2 <20 mIU / mL) and presence of vasomotor and/or menopausal symptoms (moderate to severe);
* no systemic disease (Diabetes, hypertension, hyperlipidemia, ischemic heart disease), or no infectious disease in the past 2 weeks;
* not taking any hormone therapy or medication for at least 2 months;
* no contraindications for hormone therapy in routine menopause evaluation;
* Willingness to take hormone therapy
* No smoking.

Exclusion Criteria:

* Any systemic disease (DM, HT, hyperlipidemia, ischemic heart disease) presence
* Smoking
* Contraindications for hormone therapy
* Failure to follow-up
* Inability to complete three months of hormone therapy
* Stopping hormone therapy due to vaginal bleeding during hormone therapy

Ages: 45 Years to 55 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — The treatment of menopause and hormone happens only in female sex.
Study Population: A total of cases, whose hormone therapy was planned due to menopausal symptoms in the menopause unit of our clinic, were evaluated in terms of admission, and non-acceptance criteria, during the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2008-08-30 (Actual)

PRIMARY OUTCOMES:
Blood was drawn for basal CRP from all patients | 12 months
  The patients who were evaluated for the Blatt-Kupperman index and MENQOL questionnaire were given three months of treatment to the patient, which included 1.03 mg , Estradiol hemihydrate and 0.5 mg Norethindrone acetate